CLINICAL TRIAL: NCT02667496
Title: A Study Examining the Safety and Activity of Innate Immune System Stimulation With Leukine® (Sargramostim) to Reduce Brain Amyloid Load in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease
Brief Title: Safety Study of Sargramostim in Treating Patients With Mild Cognitive Impairment Due to Alzheimer's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Sanofi (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT14019; U1111-1163-0793 (Other: UTN); 1UF1AG046143 (NIH)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Dementia Alzheimer's Type
MeSH Terms: conditions — Alzheimer Disease | interventions — sargramostim; florbetapir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leukine (Experimental): Administered SC in treatment cycles up to 24 weeks
  Florbetapir administered for PET scans to examine baseline brain imaging pathology and changes on treatment.
  Interventions: Drug: Sargramostim GZ402664; Drug: Florbetapir F18
- Placebo (Placebo Comparator): Administered SC in treatment cycles up to 24 weeks
  Florbetapir administered for PET scans to examine baseline brain imaging pathology and changes on treatment.
  Interventions: Drug: Placebo; Drug: Florbetapir F18

INTERVENTIONS:
Drug: Sargramostim GZ402664 — Pharmaceutical form:solution Route of administration: subcutaneous
  Other Names: Leukine
  Arms: Leukine
Drug: Placebo — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Placebo
Drug: Florbetapir F18 — Pharmaceutical form:solution Route of administration: intravenous

SUMMARY:
Primary Objective:

To compare the effect of repeat doses of Leukine to placebo administered subcutaneously (SC) on established cortical amyloid load in patients with mild cognitive impairment (MCI) due to Alzheimer's disease (AD).

Secondary Objective:

* To evaluate safety and tolerability of Leukine versus placebo.
* To explore the effect of Leukine versus placebo on cognitive performance.
* To collect biospecimens for future biomarker research.

DETAILED DESCRIPTION:
The total duration of study period per patient is up to 28 weeks.

ELIGIBILITY:
Inclusion criteria:

* Men and women ≥40 years and ≤80 years with a diagnosis of MCI due to AD according to the National Institutes of Aging Alzheimer's Association (NIA-AA) criteria (intermediate or high likelihood) with sporadic or familial inheritance pattern. Mild cognitive impairment AD is defined as:
* Evidence of concern about change in cognition, in comparison with person's previous level (subjective memory complaint/decline during the past year for more than 6 months and/or confirmed by informant and/or clinician), and
* Objective impairment of memory function documented by an error score on the delayed recall section of the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) ≥1.5 standard deviations (SD) from the age-stratified mean; ie,
* Age 55-69 years: ≥6 errors
* Age 70-74 years: ≥7 errors
* Age 75+ years: ≥8 errors
* But no definite impairment(s) in activities of daily living (ADLs), in the Investigator's view as assessed by the Alzheimer's Disease Cooperative Study (ADCS) ADL adapted to MCI, and
* Evidence of elevated cortical amyloid by positron emission tomography (PET) using florbetapir F18 (Amyvid) (a positive scan) by qualitative assessment according to the product label.
* Have a dedicated partner/caregiver informant who can assist the patient with the study procedures and administration of study medication, and is in the company of the patient at least 12 hours a week.
* Willing and able to provide signed informed consent.

Exclusion criteria:

* Any technical/administrative reason that makes it impossible to randomize the patient in the study.
* Prior treatment with an investigational anti-amyloid therapy.
* Contraindication for lumbar puncture, or contraindication or inability to complete magnetic resonance imaging (MRI) or having past or planned exposure to ionizing radiation that would, together with the radiation resulting from the administrations of the PET tracer used in this study, exceed applicable institutional, local, or national recommendations for annual or lifetime exposure.
* Modified Hachinski Ischemic Score >4.
* Other neurological or psychiatric condition (other than AD) which can impair cognition; or, computerized tomography (CT)/MRI evidence of potentially significant intracranial abnormalities not related to AD (eg, evidence of major stroke or lacune in an area critical to cognition, infections, cancer, hydrocephalus, multiple sclerosis etc.); or abnormal cerebrospinal fluid (CSF) not consistent with AD.
* MRI evidence of >4 microhemorrhages: patients who may be prone to spontaneous amyloid-related imaging abnormalities (ARIA-H) and/or may be more susceptible to adverse effects of the ARIA-H.
* Untreated or unstable medical condition that could interfere with the study assessments in the opinion of the Investigator or may require immune-stimulating, immune-suppressive, or immune-modulating treatment(s) during the conduct of the study; eg, immunoglobulin, therapeutic vaccines, cytokines, anti-cytokine monoclonal antibodies. History of asplenia, hyposplenia, or splenectomy (whatever the surgical reasons).
* Current mood or anxiety disorder, and/or a psychotic disorder, and/or a substance-related disorder according to Diagnostic and Statistical Manual of Psychiatric Disorders, Edition IV, text revision (DSM-IV-TR) or DSM-V; or considered suicidal or shows suicidal ideation as assessed by the Investigator.
* Laboratory abnormalities indicative of an untreated medical or hematologic condition that could increase risk or interfere with study assessments including untreated hypo- or hyperthyroidism, vitamin B12 deficiency, hyperleukocytic syndrome (including but not restricted to chronic myelogenous leukemia, Hodgkin and non-Hodgkin lymphoma), monoclonal gammopathy, and thrombocythemia.
* Known renal dysfunction or serum creatinine >150 µmol/L.
* Known hepatic dysfunction (apart from Gilbert's syndrome) or serum alanine aminotransferase (ALT) ≥3 times the upper limit of normal (ULN).
* Pregnant or breastfeeding woman.
* Presence or history of drug hypersensitivity; or known hypersensitivity to sargramostim, yeast-derived products, any other component of the product, or benzyl alcohol (present in bacteriostatic water or saline for infusion).
* Evidence of fluid retention (clinical or radiological), respiratory symptoms (eg, dyspnea), cardiovascular symptoms or electrocardiographic evidence of cardiac disease which warrant therapeutic intervention (eg, supraventricular arrhythmia).
* History of deep vein thrombosis (DVT) or pulmonary embolism or familial predisposition for DVT or pulmonary embolism.
* Women and female partners of childbearing potential and not protected by highly effective contraceptive methods of birth control (ie, oral or depot contraceptives or intrauterine device [IUD] or subject was surgically sterilized) and/or unwilling or unable to be tested for pregnancy; or are pregnant or lactating.
* Recipient of an investigational drug within prior 60 days, or within 5 times the elimination half-life of that drug, whichever is the longest.
* History of latex allergy or yeast allergy.
* Any patient who:
* Is likely to be noncompliant, leave the area, or separate from the designated caregiver/informant for more than 3 days during the study,
* Unable to cooperate because of a language problem or poor mental development,
* Oversees or implements any aspect of the study, or
* Is employed by Sanofi or its affiliates or subsidiaries (eg, Genzyme, Sanofi-Pasteur, Merial).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in standardized uptake value ratio as measured by PET using florbetapir F18 (Amyvid) | From baseline to Week 24

SECONDARY OUTCOMES:
Number of patients experiencing treatment-emergent adverse events (TEAEs) | Week 24
Change from baseline in CSF analysis | Prior to first injection on Day 1 to serve as a baseline for any necessary follow-up, and optional assessment at Day 155
MRI to assess for emergence of amyloid related imaging abnormalities (ARIA) | At Screening and Days 43, 85, and 155
Measurement of antidrug antibody levels | At Days 1, 29, 57, 85, and 155

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 840001, Houston, Texas, United States